CLINICAL TRIAL: NCT04430764
Title: The Effect of Smoking and Non-surgical Periodontal Treatment on Gingival Crevicular Fluid Cyclophilin A and EMMPRIN Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Oya Turkoglu, Professor, Ege University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014/Diş/019
Record Dates: First submitted 2020-06-09; First posted 2020-06-12 (Actual); Last update posted 2020-06-12 (Actual); Status verified 2020-06

CONDITIONS: Smoking; Periodontitis; Non-surgical Periodontal Treatment
MeSH Terms: conditions — Smoking; Periodontitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- smoker (Experimental)
  Interventions: Procedure: non-surgical periodontal treatment
- non-smoker (Active Comparator)
  Interventions: Procedure: non-surgical periodontal treatment

INTERVENTIONS:
Procedure: non-surgical periodontal treatment — Non-surgical periodontal treatment program was as following: First, motivation and oral hygiene instructions were given to all participants with periodontitis. The modified-Bass tooth brushing technique with a given dentifrice and toothbrush twice a day, and dental flossing/ interdental brushing once a day was advised to all patients with periodontitis. Second, scaling using an ultrasonic device and root planning by hand instruments under local anesthesia was performed.

SUMMARY:
This study aimed to investigate the effect of smoking and non-surgical periodontal treatment on gingival crevicular fluid CyPA and EMMPRIN levels in patients with periodontitis. Twenty-eight patients with periodontitis (14 non-smoker and 14 smoker) and 30 control subjects (15 non-smoker and 15 smoker) were included into the study. Non-surgical periodontal treatment was applied to all periodontitis patients. Periodontal parameters and GCF CyPA and EMMPRIN levels were evaluated during 3 months following non-surgical periodontal treatment. GCF CyPA and EMMPRIN levels were analyzed by ELISA.

ELIGIBILITY:
Inclusion Criteria:

* generalized periodontitis with stage III-IV & Grade B
* no systemic and periodontal diseases
* smokers (minimum 10 cigarettes per day for at least ten years)
* non-smokers (never smoked)

Exclusion Criteria:

* Systemic diseases
* Infectious diseases
* Pregnancy or lactating
* Having periodontal treatment during the last 6 months
* Having antibiotic treatment within the past 3 months
* Former smokers

Ages: 29 Years to 61 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Change in gingival crevicular fluid CypA total amounts | Baseline, 1 week, 1., 3. months
  GCF CyPA levels were analyzed by ELISA
Change in gingival crevicular fluid EMMPRIN total amounts | Baseline, 1 week, 1., 3. months
  GCF EMMPRIN levels were analyzed by ELISA

SECONDARY OUTCOMES:
Change in probing depth | Baseline, 1., 3. months
  Probing depth was measured with Williams periodontal probe.
Change in bleeding on probing | Baseline, 1., 3. months
  Bleeding on probing was evaluated the presence or absense following bleeding upon probing.

IPD SHARING:
Plan to Share IPD: Undecided